CLINICAL TRIAL: NCT07104227
Title: Effects of Body Mechanics Training on Shoulder-back Pain and Breastfeeding Ergonomics for Breastfeeding Mothers
Brief Title: Effects of Body Mechanics Training on Shoulder-Back Pain and Breastfeeding Ergonomics in Breastfeeding Mothers
Acronym: RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, AYSUN EKŞİOĞLU, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SUMEYYE BALCI; ege (Other: ege)
Record Dates: First submitted 2025-07-24; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Shoulder Pain Back Pain Postpartum Period; Back Pain; Postpartum Period
Keywords: breastfeeding; ergonomics; musculoskeletal pain
MeSH Terms: conditions — Back Pain; Breast Feeding; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Randomization: The "Demographic and Health Data Form" will be applied to the participants by the researcher responsible for randomization, and the information obtained will be kept in consecutively numbered, closed, opaque envelopes. The block randomization method will be used to divide the participants into intervention and control groups. In order to ensure balance in important demographic and health-related variables, the participants will be randomized by stratifying them according to age.
  The person responsible for collecting the study data will be unaware of the randomization process until the researcher responsible for randomization reports the results.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): After the initial data collection, the breastfeeding behaviors of the mothers in the intervention group will be observed. Then, the mothers will be given training on ergonomic breastfeeding, correct breastfeeding positions and body mechanics to strengthen the musculoskeletal system during the breastfeeding process. Then, a booklet showing the content of this training and protective movements will be shared with the mothers. Before the mothers are discharged, their breastfeeding status and pain levels will be assessed. An interview-monitoring plan will be created with the mother, stating that the follow-up data of the intervention group will be collected by telephone interview method. The mothers in the intervention group will be called at 6 weeks and 3 months after birth and their back and neck pain will be assessed.
  Interventions: Behavioral: body mechanics training; Other: to inform
- control group (Sham Comparator): The mothers in the control group will benefit from the information and support services provided by the breastfeeding consultant midwife within the scope of the hospital's routine care services. In addition, a brochure will be prepared for these mothers on the correct posture and breastfeeding positions to be considered during the breastfeeding period and will be given to them. An interview-monitoring plan will be created with the mother, stating that the follow-up data of the control group will be collected by telephone interview method. The mothers in the control group will be called simultaneously with the intervention group at the 6th week and 3rd month after birth to evaluate their back and neck pain.
  Interventions: Other: to inform

INTERVENTIONS:
Behavioral: body mechanics training — Randomization: The "Demographic and Health Data Form" will be applied to the participants by the researcher responsible for randomization, and the information obtained will be kept in consecutively numbered, closed, opaque envelopes. The block randomization method will be used when dividing the participants into intervention and control groups. In order to ensure balance in important demographic and health-related variables, the participants will be randomized by stratifying them according to age. The person responsible for collecting the study data will be unaware of the randomization process until the researcher responsible for randomization reports the results. Intervention group: After the initial data collection, the breastfeeding behaviors of the mothers in the intervention group will be observed. Then, the mothers will be given training on ergonomic breastfeeding, correct breastfeeding positions and body mechanics to strengthen the musculoskeletal system during the breas
  Arms: intervention group
Other: to inform — Kontrol grubundaki anneler, hastanenin rutin bakım hizmetleri kapsamında emzirme danışmanı ebe tarafından verilen bilgilendirme ve destek hizmetlerinden yararlanacaklardır. Ayrıca bu anneler için emzirme döneminde doğru duruş ve emzirme pozisyonlarında dikkat edilmesi gereken durumlar konusunda bir broşür hazırlanacak ve kendilerine verilecektir. Kontrol grubunun izlem verilerinin telefon görüşmesi yöntemi ile toplanacağı belirtilerek bir görüşme-izlem planı anne ile birlikte oluşturulacaktır. Kontrol grubundaki anneler müdahale grubu ile eşzamanlı olarak doğum sonu 6. Hafta ve 3.aylarda aranarak sırt ve boyun ağrıları değerlendirilecektir.

SUMMARY:
The research will be conducted as a randomized controlled trial and mothers in the intervention group will receive training on posture correction,breastfeeding positions, and shoulder and back muscle strengthening movements. If you agree to participate in this study, you will first be asked to fill out a form regarding your demographic information and health history.Then, the following scales will be applied to evaluate breastfeeding ergonomics, shoulder-back pain, and musculoskeletal system functions:Demographic and Health Data Form, Breastfeeding Ergonomics Scale, Visual Analog Scale (VAS) for Pain Assessment,Low Back Pain Function Scale, and Neck Disability Indicator Questionnaire. Mothers in the intervention group will receive training on body mechanics including posture awareness,breastfeeding positions, and shoulder and back muscle strengthening movements.The training will be conducted in the hospital and at 6 weeks and 3 months after discharge

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of body mechanics training on shoulder-back pain and breastfeeding ergonomics for breastfeeding mothers. The study is a randomized controlled intervention study. The study will be conducted in the postpartum ward of Ege University Medical Faculty Hospital. The required sample size for this study was calculated using a priori power analysis using the G*Power 3.1 program. In the calculation, a minimum of 94 people were calculated as 47 for the intervention group and 47 for the control group for a 95% confidence interval and 80% power. The study will be applied to breastfeeding mothers who have given birth vaginally; women who have given birth by cesarean section will not be included. The initial data will be collected face-to-face. Breastfeeding status and pain levels will be evaluated before the mothers are discharged. It will be stated that the follow-up data of the intervention group will be collected via telephone interview and an interview-monitoring plan will be created together with the mother. The mothers in the intervention group will be called at 6 weeks and 3 months postpartum to evaluate their back and neck pain and breastfeeding ergonomics. The mothers in the control group will be called simultaneously with the intervention group at 6 weeks and 3 months postpartum to evaluate their back and neck pain. "Demographic and Health Data Form", "Breastfeeding Ergonomics Scale", "Visual Analog Scale" for pain assessment, Low Back Pain Function Scale, and neck disability questionnaire form will be used to collect data. After the research data are obtained, the data will be analyzed using SPSS 25.0 (Statistical, Package for. Social Sciences) program. Follow-up findings of the intervention and control groups; Analysis of Variance (ANOVA) and ANCOVA will be applied to measurements with normal distribution in at least three independent group comparisons (within groups), and Kruskal Wallis analysis will be applied to measurements that do not have a normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* Mother should be 18 years of age or older
* Have given birth vaginally
* Mother should be breastfeeding
* Have good general physical health (no health problems),
* Have no physical disabilities
* Have no chronic disease (no circulatory, respiratory, endocrine, etc.)
* Have not received any physical therapy or manual therapy in the last 6 months
* Have no history of chronic pain related to the musculoskeletal system (fibromyalgia, chronic low back or neck pain, etc.)
* Have a BMI between 18.5 and 24.9
* Have a healthy newborn
* Plan to continue breastfeeding during the study period
* Have no past or current health problems that may affect breastfeeding (breast surgery, use of medications that may affect breastfeeding, etc.)
* The most less than primary level education

Exclusion Criteria:

* Mothers with any medical history
* Mothers with postural problems (previously diagnosed serious postural disorders such as scoliosis, kyphosis or lordosis)
* Having an orthopedic or neurological disorder diagnosed before or during pregnancy (herniated disc, nerve compression)
* Having had a Caesarean section
* Mothers not wanting to breastfeed
* Mothers not wanting to participate in the study
* Situations where the mother and baby must be separated
* Mothers planning to start a different exercise program during the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — She must be a woman because she has given birth and is breastfeeding.
Enrollment: 94 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Shoulder and Upper Back Pain Intensity in Breastfeeding Mothers Measured by Visual Analog Scale (VAS) | Baseline (hospital discharge), 6 weeks postpartum, 3 months postpartum
  Pain intensity will be measured using the Visual Analog Scale (VAS) in both the intervention and control groups. VAS is a 10-cm horizontal line where 0 indicates "no pain" and 10 indicates "worst pain imaginable." Scores will be recorded at baseline (hospital discharge), at 6 weeks, and at 3 months postpartum. The primary outcome is the difference in VAS scores between groups over time.
Change in Breastfeeding Ergonomics Score Measured by the Breastfeeding Ergonomics Assessment Scale (BEAS) | Baseline, 6 weeks, 3 months postpartum
  The Breastfeeding Ergonomics Assessment Scale (BEAS), developed by Ekşioğlu & Balcı (2024), consists of 14 items with a total score ranging from 14 to 42. Higher scores indicate greater ergonomic risk during breastfeeding. The scale will be administered at baseline (hospital discharge), at 6 weeks, and 3 months postpartum. The outcome is the change in BEAS score over time between the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: AYSUN EKŞİOĞLU, Associate Professor, Study Director — Ege University
Locations (1):
- Ege University, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We think that the study will be interpreted better.

REFERENCES:
- [Background] Afshariani R, Kiani M, Zamanian Z. The influence of ergonomic breastfeeding training on some health parameters in infants and mothers: a randomized controlled trial. Arch Public Health. 2019 Nov 11;77:47. doi: 10.1186/s13690-019-0373-x. eCollection 2019. PMID 31737269